CLINICAL TRIAL: NCT05521698
Title: A Randomized Trial of Apalutamide in Non-Muscle Invasive Bladder Cancer
Brief Title: Study to Determine Possible Effects of Apalutamide, Compared to Placebo, on EGFR Expression in Patients With Non-muscle Invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCI-2022-06871; NCI-2022-06871 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pending12 (Other: University of Wisconsin Carbone Cancer Center - University Hospital); INT22-09-01 (Other: DCP); P30CA014520 (NIH); UG1CA242635 (NIH)
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Non-Muscle Invasive Bladder Urothelial Carcinoma; Recurrent Non-Muscle Invasive Bladder Urothelial Carcinoma
MeSH Terms: interventions — apalutamide; Biopsy; Specimen Handling; Transurethral Resection of Bladder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants and the study team will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (apalutamide,TURBT) (Experimental): Patients receive apalutamide PO QD on days 1-21. Patients undergo TURBT on day 21. Up to 28 days of apalutamide prior to TURBT is permitted in the absence of unacceptable toxicity. Patients undergo blood and urine sample collection throughout the study. Patients may optionally undergo tumor biopsy at baseline.
  Interventions: Drug: Apalutamide; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Procedure: Transurethral Resection of Bladder Tumor
- Arm 2 (placebo, TURBT) (Placebo Comparator): Patients receive placebo PO QD on days 1-21. Patients undergo TURBT on day 21. Up to 28 days of placebo prior to TURBT is permitted in the absence of unacceptable toxicity. Patients undergo blood and urine sample collection throughout the study. Patients may optionally undergo tumor biopsy at baseline.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration; Procedure: Transurethral Resection of Bladder Tumor

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
  Arms: Arm 1 (apalutamide,TURBT)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Placebo Administration — Given PO
  Arms: Arm 2 (placebo, TURBT)
Other: Questionnaire Administration — Ancillary studies
Procedure: Transurethral Resection of Bladder Tumor — Undergo TURBT
  Other Names: Transurethral resection (TURBT); TURBT

SUMMARY:
This phase I trial evaluates the effects of apalutamide, compared to placebo, on epidermal growth factor receptor (EGFR) protein expression in patients with non-muscle invasive bladder cancer. Apalutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of tumor cells. Previous studies have suggested that expression of a protein called EGFR on tumor cells is related to bladder cancer disease progression. This trial may help doctors evaluate if apalutamide has any effect on EGFR expression in patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare epidermal growth factor receptor (EGFR) messenger ribonucleic acid (mRNA) expression measured by reverse transcriptase polymerase chain reaction (rt-PCR) in normal appearing urothelium adjacent to tumor (measured as a ratio relative to urothelium and lamina-propria specific markers) in participants treated with anti-androgen therapy versus (vs.) participants given placebo.

SECONDARY OBJECTIVES:

I. To determine effect of apalutamide on EGFR expression (by rtPCR) in the subgroup of patients whose normal appearing urothelium adjacent to tumor expresses the androgen receptor (AR) (at least "1" by immunohistochemistry [IHC] score).

II. To correlate AR expression in adjacent urothelium (by IHC score) with EGFR expression by rtPCR in participants randomized to apalutamide versus placebo.

III. Comparison of toxicity in participants randomized to apalutamide versus placebo.

EXPLORATORY OBJECTIVES:

I. Comparison of AR and EGFR (and possibly phosphorylated EGFR [pEGFR]) staining levels (low, moderate, high; by immunocytology) in pre-treatment vs. post-treatment bladder wash cytology.

II. To compare expression of direct androgen response gene (ADAR)-2 measured by rtPCR in normal appearing adjacent (to tumor) urothelium that does and does not express AR (by IHC), in participants randomized to apalutamide versus placebo.

III. Ki-67 expression (by IHC) in normal appearing urothelium adjacent to tumor in participants randomized to apalutamide versus placebo.

IV. Subgroup analysis of Ki-67 expression in the AR+ subgroup. V. Differences in expression of AR, EGFR, pEGFR, and Ki-67 (by semi-quantitative IHC) in tumor in participants randomized to apalutamide versus placebo.

VI. Comparison of demographics of two groups. VII. Change in EGFR expression by rt-PCR in tumor in participants randomized to apalutamide versus placebo.

VIII. Morbidities of treatment (breast tenderness, sexual or urinary side effects, seizure[s], depression, abnormal liver function tests [LFTs]).

IX. Comparison of pre vs. post intervention urinary biomarkers (CxBladderTM) in both groups, examining the 5 RNAs (by rtPCR) that make up the test, both as a group and each RNA separately.

X. Fibroblast growth factor receptor 3 (FGFR3) mutation analysis in deoxyribonucleic acid (DNA) extracted from formalin fixed paraffin embedded (FFPE) blocks from neighboring normal urothelium and tumor tissue in participants randomized to apalutamide versus placebo.

XI. Define changes in the tumor immune microenvironment pre- and post-apalutamide through liquid biopsies of blood and urine using high-dimensional flow cytometry.

XII. Analyze tumor (biopsy specimen) immune microenvironment via multiplex immunofluorescence and spatial transcriptomics.

XIII. Compare AR, EGFR, and pEGFR in biopsies of tumors done at index cystoscopy vs. TURBT in participants randomized to apalutamide versus placebo. (Optional) XIV. Other exploratory markers such as changes in the urinary microbiome in bladder cancer participants randomized to apalutamide versus placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive apalutamide orally (PO) once daily (QD) on days 1-21. Patients undergo TURBT on day 21. Up to 28 days of apalutamide prior to TURBT is permitted in the absence of unacceptable toxicity. Patients undergo blood and urine sample collection throughout the study. Patients may optionally undergo tumor biopsy at baseline.

ARM 2: Patients receive placebo PO QD on days 1-21. Patients undergo TURBT on day 21. Up to 28 days of placebo prior to TURBT is permitted in the absence of unacceptable toxicity. Patients undergo blood and urine sample collection throughout the study. Patients may optionally undergo tumor biopsy at baseline.

After completion of study treatment, patients are followed up 20-30 days after TURBT.

ELIGIBILITY:
Inclusion Criteria:

* Biologic male adults (>= 18 years old)

  * Note: Because no dosing or adverse event (AE) data are currently available on the use of apalutamide in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable
* Have suspected non-muscle invasive bladder carcinoma (NMIBC) on clinic-based cystoscopy or imaging as viewed by an American Urological Association (AUA) board-certified urologist
* Have had cross sectional imaging of the abdomen and pelvis (computed tomography [CT] or magnetic resonance imaging [MRI] with or without contrast) within 6 months prior to enrollment with no signs of upper tract urothelial cancer (UC), invasive, nor metastatic disease

  * Note: If adenopathy or upper tract abnormalities are identified, a negative biopsy and or ureteroscopy is required prior to enrollment
* Newly suspected, diagnosed, or occasionally recurrent bladder cancer (BC)

  * Note: Occasional recurrence is defined as =< 2 prior NMIBC episodes in the 18 months preceding cystoscopy where the index tumor was identified
* Participants with single and multiple tumor lesions
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Total bilirubin =< 1.5 x institutional upper limit of normal (note: in participants with Gilbert's syndrome, if total bilirubin is > 1.5 x upper limit of normal, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x upper limit of normal, participants may be eligible)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2 × institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2 × institutional upper limit of normal
* Urine Culture < 50,000 colonies/cc of 1 or more organisms (if found and treated and a confirmed negative culture obtained off antibiotics before study drug is started, they will be eligible)
* Serum Testosterone >= 300 ng/dL
* Thyroid stimulating hormone (TSH) within institutional normal
* White blood cell count (WBC) >= 0.5 × institutional lower limit of normal
* The effects of apalutamide on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, men who are having sex must wear a condom when engaging in any activity that allows for passage of ejaculate to another person throughout the course of the study and 90 days after receiving last dose of study intervention. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak. Additionally, men must agree to not donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study intervention
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had a previous exposure to sex hormone (e.g., exogenous androgens) or anti-androgenic therapies (e.g., luteinizing hormone-releasing hormone [LHRH] agonists, LHRH antagonists, 5 alpha reductase-inhibitors, abiraterone or other anti-androgens) within 6 months of accrual
* Participants who are taking the following medications that increase seizure risks: (e.g., clozapine, olanzapine, risperidone, ziprasidone), phenothiazine, antipsychotics (e.g., chlorpromazine, mesoridazine, thioridazine), bupropion, lithium, meperidine, pethidine, phenothiazine and tricyclic antidepressants (e.g., amitriptyline, desipramine, doxepin, imipramine, maprotiline), mirtazapine, selective serotonin reuptake inhibitors (e.g., escitalopram, citalopram, fluoxetine), serotonin norepinephrine reuptake inhibitors (e.g., venlafaxine, desvenlafaxine, levomilnacipran), stimulants (e.g., amphetamines, methylphenidate), monoamine oxidase inhibitors (e.g., phenelzine, selegiline)
* Participants taking any form of anticoagulation (e.g., heparin, warfarin, lovenox, apixaban, rivaroxaban, dabigatran, edoxaban, betrixaban)
* Concurrent use of drugs in category X drug interactions with apalutamide
* Participants receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to apalutamide
* History of prior or concurrent muscle invading UC, or concurrent prostatic urethral, urethral, or upper tract UC or non-urothelial bladder cancer
* History of radiation therapy to the pelvis, prostate or prostatic bed, or rectum
* Any condition (uncontrolled intercurrent illness, psychiatric illness, or social situation) for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* History of seizures or central nervous system (CNS) metastasis or any condition that in the opinion of the investigator may predispose to seizure or treatment with drugs known to lower the seizure threshold within 4 weeks prior to enrollment in the study
* Participants with severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, uncontrolled hypertension, long QT, arterial or venous thromboembolic events (eg pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias
* In the opinion of the investigator, participant has uncontrolled hypertension, high cholesterol, or diabetes
* Allergy or hypersensitivity to apalutamide, or excipients, unable or unwilling to take antiandrogen therapy (ADT)
* Plans to father a child while enrolled in this study or within 12 weeks after the last dose of study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Average Epidermal Growth Factor Receptor (EGFR) expression level | Up to 28 days
  Will be analyzed as a continuous variable. A two-sample t-test will be conducted to test whether there are significant differences of the log-transformed EGFR expression level (measured by reverse transcriptase polymerase chain reaction [rtPCR]) in normal appearing urothelium adjacent to tumor in participants treated with anti-androgen therapy versus (vs.) placebo participants. In case the normality assumption of the two-sample t-test does not hold, Wilcoxon rank-sum test will be performed as a sensitivity analysis. Considering androgen receptor (AR) status can be a treatment effect modifier, a regression analysis will also be performed with the log-transformed EGFR expression level as the outcome and treatment status (apalutamide or placebo), AR status, and treatment-AR interaction as the predictors.

SECONDARY OUTCOMES:
Effect of apalutamide on EGFR expression | Up to 28 days
  A two-sample Wilcoxon rank-sum test will be conducted to compare the difference of EGFR expression in AR positive participants treated with and without apalutamide.
AR expression in adjacent urothelium | Up to 28 days
  Will evaluate the correlation between AR expression in adjacent urothelium with EGFR expression. Pearson correlation and Spearman's rank correlation will be calculated between the AR expression and EGFR expression.
Toxicity of treatment | Up to 28 days
  Toxicity of treatment may include breast tenderness, sexual or urinary side effects, seizure(s), depression, abnormal liver function tests. Descriptive statistics will be provided for these outcomes.

OTHER OUTCOMES:
AR and EGFR (and possibly phosphorylated EGFR [pEGFR]) staining levels | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Expression of direct androgen response gene (ADAR)-2 | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Ki-67 expression | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Ki-67 expression in the AR+ subgroup | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Differences in expression of AR, EGFR, pEGFR, and Ki-67 | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Demographics of two groups | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Change in EGFR expression in tumor from participants randomized to apalutamide versus placebo | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Morbidities of treatment | Up to 28 days
  Morbidities of treatment may include breast tenderness, sexual or urinary side effects, seizure(s), depression, abnormal LFTs. Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Pre vs. post intervention urinary biomarkers | Up to 28 days
  Comparison of pre vs. post intervention urinary biomarkers (CxBladderTM) in both groups, examining the 5 ribonucleic acids (RNAs) (by rtPCR) that make up the test, both as a group and each RNA separately. Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Analysis of fibroblast growth factor receptor 3 (FGFR3) in deoxyribonucleic acid (DNA) | Up to 28 days
  Extracted from fixed paraffin embedded (FFPE) blocks from neighboring normal urothelium and tumor tissue in participants treated with or without apalutamide. Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
Changes in the tumor immune microenvironment pre- and post-apalutamide | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions.
Analysis of tumor (biopsy specimen) infiltrating CD8+ T-cells | Up to 28 days
  The tumor immune microenvironment will be analyzed via multiplex immunofluorescence and spatial transcriptomics. Assessments will include CD8+ T-cell functional markers: TCF1/Tcf7 of CD44+, CD62L, PD-1, TIM3 and SLAMF6. Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.
AR, EGFR, and pEGFR in biopsies of tumors | At index cystoscopy and TURBT
  Optional biopsy tissue will be used to compare AR, EGFR, and pEGFR in biopsies of tumors done at index cystoscopy vs. transurethral resection of bladder tumor in participants randomized to apalutamide versus placebo.
Exploratory markers | Up to 28 days
  Will be summarized by descriptive statistics such as rates and proportions and compared between placebo and apalutamide using nonparametric tests such as the Kruskal-Wallis test.

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Messing, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - University of Arizona Cancer Center - Prevention Research Clinic, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - National Cancer Institute Urologic Oncology Branch, Bethesda, Maryland
  - University of Rochester, Rochester, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm